CLINICAL TRIAL: NCT07328412
Title: Aromatherapy to Address Psychological Distress in Emergency Department Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Peter R Chai MD, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025P002810
Record Dates: First submitted 2025-12-01; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Aromatherapy; Anxiety; Stress; Emergency Department
MeSH Terms: conditions — Anxiety Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy Group (Experimental): Participants will receive a lavender-scented tube to inhale for 5 minutes.
  Interventions: Other: Lavender Aromatherapy
- Control Group (Active Comparator): Participants will receive an unscented tube to inhale for 5 minutes.
  Interventions: Other: Unscented Aromatherapy

INTERVENTIONS:
Other: Lavender Aromatherapy — A diffuser tube containing a cotton wick infused with 5 drops of lavender essential oil.
  Arms: Aromatherapy Group
Other: Unscented Aromatherapy — A diffuser tube containing a cotton wick saturated with 10 drops of water.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to understand the feasibility and acceptability of a brief aromatherapy session for reducing stress, anxiety, and improving patient satisfaction among emergency department patients. The main question the study aims to answer is: Is the intervention acceptable and feasible? Participants in the intervention group will receive a lavender-scented tube and smell it for about 5 minutes. Participants in the control group will receive an unscented tube and follow the same instructions.

DETAILED DESCRIPTION:
Stress and anxiety are frequently experienced by patients during emergency department (ED) visits, often due to diagnostic uncertainty, prolonged wait times, and environmental factors such as noise and bright lighting. These psychological stressors can trigger physiological responses, including elevated cortisol levels, increased blood pressure, and disrupted sleep, which may negatively impact patients' experiences and overall health outcomes. Aromatherapy has emerged as a promising non-pharmacologic intervention for reducing stress and anxiety in various settings.

This pilot randomized controlled trial will be conducted to assess the feasibility and acceptability of a brief aromatherapy session for ED patients. Research staff will pre-screen potential participants admitted to the ED Observation Unit at Brigham and Women's Hospital (BWH) using information from the electronic medical record. After obtaining approval from the treating medical team, staff will approach and invite potential participants to participate in the study. Once consented and screened eligible, participants will complete a baseline assessment and be randomized in a 1:1 ratio to either the aromatherapy group or the control group. Participants in the aromatherapy group will receive a lavender-scented tube and be instructed to inhale it for about 5 minutes. Participants in the control group will receive an unscented tube and follow the same instructions. After the session, participants will complete a post-experiment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Admitted to the BWH Emergency Department (ED) Observation Unit
* Able to provide written informed consent
* Willing to participate in a 1-hour aromatherapy session

Exclusion Criteria:

* Acutely ill and unable to be approached for research, as determined by the treating medical team and/or physician investigator
* Active gastrointestinal problems at the time of enrollment (e.g., nausea, vomiting, abdominal cramping, diarrhea), as determined by the treating team and/or physician investigator.
* Pregnancy or breastfeeding
* Current or planned treatment using sedating medications
* History of, or current presentation with, significant cognitive impairment or acute delirium that would preclude informed consent or participation
* Currently receiving supplemental oxygen
* Acute exacerbation of asthma or COPD
* Admission for an acute upper or lower respiratory tract illness (e.g., pneumonia, bronchitis, influenza, COVID-19)
* Known allergy or sensitivity to lavender
* Documented history of anosmia (loss of smell)
* Documented hypotension during current ED presentation, defined as systolic blood pressure <90 mmHg
* Assigned clinical staff (physician, nurse, or other healthcare provider) with fragrance sensitivity prior to consent
* Concurrent enrollment in another interventional drug or behavioral trial
* Any condition that, in the judgment of the treating team or physician investigator, would make study participation unsafe or inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention via AIM | day 1
  Acceptability will be assessed via the Acceptability of Intervention Measure (AIM). AIM is a 4-item Likert agreeability scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated, resulting in a continuous score with higher scores indicating greater intervention acceptability.
Usability of intervention via SUS | day 1
  Usability will be assessed via an adapted, validated 2-item version of the System Usability Scale (SUS). Each item is rated on a 5-point Likert scale from 1 (Strongly disagree) to 5 (Strongly agree). The mean score of each item will be calculated and entered into a validated regression equation to estimate the full SUS score, which ranges from 0 to 100, with higher scores indicating greater usability.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chai, MD, MMS, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No